CLINICAL TRIAL: NCT03222219
Title: Influence of the Implant Insertion Torque on the Primary Stability of Tapered Dental Implants With Deep Spires
Brief Title: Implant Insertion Torque and Primary Stability
Acronym: TorqueISQ
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the Academy, International Piezosurgery Academy
Other Study IDs: TorqueISQ
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: DENTAL IMPLANTATION
Keywords: dental implant insertional torque stability
MeSH Terms: interventions — Torque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low implant stability quotient: dental implant insertion with low torque values
  Interventions: Procedure: dental implant insertion
- medium implant stability quotient: dental implant insertion with medium torque values
  Interventions: Procedure: dental implant insertion
- high implant stability quotient: dental implant insertion with high torque values
  Interventions: Procedure: dental implant insertion

INTERVENTIONS:
Procedure: dental implant insertion — the registration of the torque values is discriminant for the group assignment after dental implant insertion
  Other Names: torque and stability quotient

SUMMARY:
The objective of this observational study is to evaluate the primary stability of dental implants. Clinical insertion torque data with the Implant Stability Quotient will be correlated.

DETAILED DESCRIPTION:
In the healing of long bone fractures, the absence of movement between the two parts of the fracture is essential for good healing: the movement, even at the micrometric level, can generate stress and tensions that prevent bone apposition in the gap. Even the primary stability of a dental implant is one of the main preconditions for osseointegration: in fact, during healing, micromovies that exceed the threshold of 100-150 microns can stimulate the growth of fibrous tissue in the bone to implant interface, leading to the failure of the procedure.

It is also known that primary implant stability tends to decrease in the first weeks after placement due to inflammatory response due to surgical trauma before rising when bone recoating phenomena begin to prevail over reabsorption. Attention to implant stability is a crucial factor, especially in cases where immediate or early loading procedures are in place: system stress during chewing or simply related to tongue, cheeks or lips movements can result in micromovements that may lead to the failure of the procedure.

With these assumptions, it is evident that a tool that allows the clinician to have a reliable evaluation of implant stability is the most important one: currently in use are the measurement of the insertion torque of the implant and the resonance frequency analysis. The insertion torque can be defined as the measurement of the resistance that the system encounters during its advancement in the apical direction by means of a rotating movement on its axis. Resonance frequency analysis is a not invasive method that evaluates rigidity of the bone system by measuring the size of the implant movement under a lateral force. High insertion torques have been proposed as a first rate technique to achieve a great implant stability, especially in cases to be treated with immediate or early load; Other studies point out that excessive insertion torques can cause both biological problems and mechanical to the implant.

However, the relationship between insertion torque and implant stability is unclear: according to some in vitro studies, the two elements would be in direct relation, while others would be independent.

The purpose of this prospective study is to evaluate in vivo the relationship between insertion torque value and implant stability measured using resonance frequency analysis in dental implants with a deep spire conical design.

ELIGIBILITY:
Inclusion Criteria:

1. indications for insertion of dental implants, based on careful diagnosis and treatment plan;
2. presence of a residual bone crest with a height ≥ 11 mm and thickness ≥ 6 mm at the site of the implant site planned;
3. the bone crest must be intact (at least 3 months after the loss / extraction of the corresponding dental element);
4. age of the patient more than 18 years;
5. patients should be able to examine and understand the protocol of study;
6. informed consent.

Exclusion Criteria:

1. acute myocardial infarction in the last six months;
2. uncontrolled clotting disorders;
3. unmanaged diabetes (HBA1c superior than 7.5%);
4. radiotherapy in the head / neck district for the last 24 months;
5. Immune compromise (HIV infection or chemotherapy over the last 3 years);
6. active or past treatment with intravenous bisphosphonates;
7. psychological or psychiatric diseases;
8. abuse of alcohol or drug use;
9. unregulated periodontal disease;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was composed of all patients presenting for evaluation and management of any single edentulism requiring single dental implant insertion with healed bone crest and sufficient recipient bone. To be included in the study sample, patients had to present a residual crestal height more than 11 mm, wider more than 6 mm and to be 18 years or older, and able to understand and sign a written informed consent form.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
insertional torque value | during surgery
  registration of torque values with dedicated device

SECONDARY OUTCOMES:
radiographic assessment | 6 months after surgery
  intra oral radiographs are produced for crestal bone assessment
clinical assessment | 12 months after surgery
  clinical evaluation of the dental implant
implant stability quotient | during surgery
  registration of implant stability quotient with dedicated device

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Acil Y, Sievers J, Gulses A, Ayna M, Wiltfang J, Terheyden H. Correlation between resonance frequency, insertion torque and bone-implant contact in self-cutting threaded implants. Odontology. 2017 Jul;105(3):347-353. doi: 10.1007/s10266-016-0265-2. Epub 2016 Aug 18. PMID 27538921
- [Result] Santamaria-Arrieta G, Brizuela-Velasco A, Fernandez-Gonzalez FJ, Chavarri-Prado D, Chento-Valiente Y, Solaberrieta E, Dieguez-Pereira M, Vega JA, Yurrebaso-Asua J. Biomechanical evaluation of oversized drilling technique on primary implant stability measured by insertion torque and resonance frequency analysis. J Clin Exp Dent. 2016 Jul 1;8(3):e307-11. doi: 10.4317/jced.52873. eCollection 2016 Jul. PMID 27398182
- [Derived] Baldi D, Lombardi T, Colombo J, Cervino G, Perinetti G, Di Lenarda R, Stacchi C. Correlation between Insertion Torque and Implant Stability Quotient in Tapered Implants with Knife-Edge Thread Design. Biomed Res Int. 2018 May 15;2018:7201093. doi: 10.1155/2018/7201093. eCollection 2018. PMID 29862286